CLINICAL TRIAL: NCT05093660
Title: Diagnostic Importance of the Circulating Human Leucine-rich α-2-glycoprotein Analysed From Blood and Saliva in Children With Acute Appendicitis
Brief Title: Diagnostic Importance of the Circulating Human Leucine-rich α-2-glycoprotein in Acute Appendicitis in Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KBC Split (Other)
Responsible Party: Principal Investigator, Goran Tintor, Plastic surgery resident, KBC Split
Other Study IDs: 2181-147/01/06/M.S.-20-02
Record Dates: First submitted 2021-09-19; First posted 2021-10-26 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with acute appendicitis: Patients with acute appendicitis, after surgery and with pathohistological specimen confirmation.
  Interventions: Diagnostic Test: Blood specimen collection; Diagnostic Test: Saliva specimen collection
- Patients without acute appendicitis: Patients without acute appendicitis, after laboratory, clinical and/or radiological exclusion of acute admittance.
  Interventions: Diagnostic Test: Blood specimen collection; Diagnostic Test: Saliva specimen collection

INTERVENTIONS:
Diagnostic Test: Blood specimen collection — Blood specimen collection for analysis of CRP (C-reactive protein), WBC (White blood cells) and LRG1 (Circulating Human Leucine-rich α-2-glycoprotein) levels
Diagnostic Test: Saliva specimen collection — Saliva specimen collection for analysis of LRG1 (Circulating Human Leucine-rich α-2-glycoprotein) levels

SUMMARY:
Acute appendicitis is a common and potentially serious medical condition which can be difficult to diagnose, especially in pediatric patients. To help recognize patients with acute appendicitis, number of laboratory and radiological test are used. Previous research has shown that Circulating Human Leucine-rich α-2-glycoprotein (LGR1) in the blood can be elevated in pediatric patients with acute appendicitis. The aim of this research is to analyse whether LGR1 levels in saliva can be used as a less invasive diagnostic method in pediatric patients with suspected acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* children with age from 5 do 17 with acute abdominal pain
* children with clinical signs of appendicitis

Exclusion Criteria:

* previous diagnosis of chronic and/or malignant disease
* children which had previous abdominal surgery
* pregnancy

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients from 5 to 17 years of age, presenting with acute abdominal pain consistent with diagnosis of acute appendicitis, to Emergency Surgery Department at the University Hospital Split.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Level of LGR1 protein in blood | 72 hours
  Levels of LGR1 protein in blood and saliva as measured by ELISA test
Level of LGR1 protein saliva | 72 hours
  Levels of LGR1 protein in saliva as measured by ELISA test

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Split, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: No